CLINICAL TRIAL: NCT05838599
Title: Combining Topical Imiquimod With Local Radiotherapy for Treatment of Mycosis Fungoides
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Xiaolong (Alan) Zhou, Principal Investigator, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AZ10312022
Record Dates: First submitted 2023-02-06; First posted 2023-05-01 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Mycosis Fungoides
MeSH Terms: conditions — Mycosis Fungoides | interventions — Imiquimod; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Topical IMQ and localized RT (Experimental): After the initial study visit, patients will immediately begin use of imiquimod cream at designated lesions (those with combined size >50cm2) nightly for 5 consecutive days a week over 6 weeks. One week into the imiquimod treatment course, radiation therapy will be administered at Northwestern Medicine by radiation oncologists familiar with MF in 2 fractions of 4 Gy (total 8 Gy) over 2 days to the same designated lesions.
  Interventions: Drug: Imiquimod; Radiation: Radiation Therapy

INTERVENTIONS:
Drug: Imiquimod — 5% cream applied topically 5 days/week for 6 weeks
Radiation: Radiation Therapy — 2 fractions of 4 Gys (total of 8 Gys) starting 1 week after Imiquimoid course over 2 days.

SUMMARY:
Mycosis fungoides (MF) is the most common subtype of cutaneous T cell lymphoma (MF) and presents as cutaneous patches, plaques, and tumors. Radiation therapy (RT) is a frequently pursued management option for CTCL, especially in patients with more advanced skin disease. Imiquimod stimulates a Th1 lymphocyte response with increased IL-2 and IFN-α, but also induces IFN-α, TNF-α, IL-1α, IL-6, and IL-8, thereby bridging both innate and adaptive immunity. Dosing of both radiotherapy (RT) and imiquimod are based on standard-of-care doses/frequencies for CTCL. The reason imiquimod topical is given for a week before giving RT is to prime innate immune activity for when RT is delivered. It is believed that this serves as an adjuvant for the CD8+ antitumor response generated by RT. The primary aim of this study is to assess the safety and efficacy of a combination local radiotherapy and topical imiquimod approach for the treatment of conventional (CD4+) MF.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have confirmed stage IA-IIB mycosis fungoides.
* Patients must be 18-90 years of age.
* Patients must have failed at least one standard therapy for MF.
* Patients must have active, but stable disease for >6 months.
* Patients must have 4 or more discrete MF lesions with at least 2 of them with minimum combined surface area of >50cm2.
* POCBP must have a negative pregnancy test prior to registration on study.
* Patients must have the ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Patients who are on current systemic or topical CTCL therapy, unless stable on the treatment for >6 months.
* Patients who have received antibiotic therapy within 4 weeks of study enrollment.
* Patients who are pregnant or nursing. Pregnant people are excluded from this study because IMQ is an agent with potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the gestational parent with IMQ, breastfeeding should be discontinued if the parent is treated with IMQ.
* Patients with psychiatric illness/social situations that would limit compliance with study requirements.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2023-07-24 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Efficacy of a combination local radiotherapy and topical imiquimod approach for the treatment of conventional (CD4+) MF as measured by mSWAT at week 8. | 8 weeks
  The primary efficacy endpoint will be skin disease response as measured by mSWAT (Modified Severity-Weighted Assessment Tool) at week 8.
Incidence of treatment-emergent adverse events (safety and tolerability) of a combination local radiotherapy and topical imiquimod approach for the treatment of conventional (CD4+) MF. | 12 weeks
  Adverse event occurrence during study.

SECONDARY OUTCOMES:
Microbiome alterations before and after treatment | 12 weeks
  To measure alterations in lesional (tumor-associated) skin, nasal, and gut microbiomes before and after combination RT/imiquimod treatment and associate these differences in microbiomes with clinical response (and any toxicity). Differences in microbiome bacterial species will be measured by alpha and beta diversity metrics. Alpha diversity quantifies within sample diversity. Beta diversity compares between sample diversity (before and after treatment).
Tumor-associated and serum immune alterations before and after treatment | 12 weeks
  To correlate quantitative changes in tumor-associated and serum immune response profiles with clinical response to RT/imiquimod treatment (and any toxicity).

CONTACTS AND LOCATIONS:
Overall Officials: Alan Zhou, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University Department of Dermatology, Chicago, Illinois, United States